CLINICAL TRIAL: NCT03139448
Title: Comparison of Oxygenation and Ventilation With a Novel Nasal Mask Versus Standard of Care During Colonoscopy: a Prospective Randomized Trial
Brief Title: Comparison of Oxygenation and Ventilation With a Novel Nasal Mask Versus Standard of Care During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Revolutionary Medical Devices, Inc. (Unknown)
Responsible Party: Principal Investigator, Koffi Michael Kla, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170488
Record Dates: First submitted 2017-05-01; First posted 2017-05-04 (Actual); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Colonoscopy; Oxygenation; Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Oxygen via nasal cannula (Standard of Care) (Active Comparator): The anesthesia provider will supply oxygen via nasal cannula at oxygen flow rates as per standard of care routine at Vanderbilt University Medical Center.
  Interventions: Device: Oxygen via nasal cannula
- Oxygen via SuperNO2VA nasal mask (Experimental): The anesthesia provider will attach the SuperNO2VA's (Revolutionary Medical, Inc) circuit port to the anesthesia machine, turn the oxygen flow rate to 10L/min, and set the APL valve to 10 cm H2O.
  Interventions: Device: Oxygen via SuperNO2VA nasal mask

INTERVENTIONS:
Device: Oxygen via nasal cannula — Oxygen will be supplied to the patient via nasal cannula according to the routine standard of care practice at Vanderbilt University Medical Center.
  Arms: Oxygen via nasal cannula (Standard of Care)
Device: Oxygen via SuperNO2VA nasal mask — The anesthesia provider will attach the SuperNO2VA's (Revolutionary Medical, Inc) circuit port to the anesthesia machine, turn the oxygen flow rate to 10L/min, and set the APL valve to 10 cm H2O.
  Arms: Oxygen via SuperNO2VA nasal mask

SUMMARY:
Nasal continuous positive airway pressure (nCPAP) has been shown to effectively relieve upper airway obstruction in patients with OSA as it creates a pneumatic stent in the hypopharynx that reduces obstruction and allows for continuous oxygenation. Nasal ventilation was also proven to be more effective than combined oral-nasal ventilation during induction of general anesthesia in adult subjects. However, it is not clear if nasal mask can be used safely for oxygenation and ventilation in patients undergoing colonoscopy.

The SuperNO2VA™ device is a new commercially available nasal mask that provides both nasal CPAP and nasal mask ventilation. The objective of this study is to compare the efficacy of oxygenation and ventilation during colonoscopy using the novel nasal mask, SuperNO2VA™, and standard care with nasal cannula.

DETAILED DESCRIPTION:
Colonoscopy has become an essential part of the patient management, especially in the field of colorectal cancer prevention. About 15 million colonoscopies were done in the United States in 2012. Data from United States and European countries suggest that the majority of investigations are performed with the aid of sedation. Since sedation can cause significant respiratory depression, resulting in hypoxia, especially in obese and elder populations who are more likely to undergo colonoscopy, usually oxygen is provided to patients via a nasal cannula to minimize the risk of hypoxia.

Nasal continuous positive airway pressure (nCPAP) has been shown to effectively relieve upper airway obstruction in patients with OSA as it creates a pneumatic stent in the hypopharynx that reduces obstruction and allows for continuous oxygenation. Nasal ventilation was also proven to be more effective than combined oral-nasal ventilation during induction of general anesthesia in adult subjects. However, it is not clear if nasal mask can be used safely for oxygenation and ventilation in patients undergoing colonoscopy.

The SuperNO2VA™ device is a new commercially available nasal mask that provides both nasal CPAP and nasal mask ventilation. The objective of this study is to compare the efficacy of oxygenation and ventilation during colonoscopy using the novel nasal mask, SuperNO2VA™, and standard care with nasal cannula.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* BMI of 30-50
* ASA 1-3 Scheduled for colonoscopy with sedation

Exclusion Criteria:

* Untreated ischemic heart disease
* Acute and chronic respiratory disorders, including COPD and asthma
* Emergent procedures
* Planned use of an invasive airway (ie: supra-glottic device, LMA, etc)
* Pregnant women
* Nasal or oral disease resulting in difficulty of either nasal breathing or mouth breathing
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koffi M Kla, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bai Y, Xu Z, Chandrashekar M, St Jacques PJ, Liang Y, Jiang Y, Kla K. Comparison of a simplified nasal continuous positive airways pressure device with nasal cannula in obese patients undergoing colonoscopy during deep sedation: A randomised clinical trial. Eur J Anaesthesiol. 2019 Sep;36(9):633-640. doi: 10.1097/EJA.0000000000001052. PMID 31313720

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxygen Via Nasal Cannula (Standard of Care) | Oxygen Via SuperNO2VA Nasal Mask
Started (All participants randomized) | 85 | 89
Intervention Started (All participants that received partial or full intervention) | 79 | 70
Completed (Participants that received a full intervention) | 73 | 63
Not Completed | 12 | 26
Not completed — Lack of Efficacy | 6 | 7
Not completed — Location of procedure changed | 2 | 8
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Screen fail | 1 | 3
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxygen Via Nasal Cannula (Standard of Care) | Oxygen Via SuperNO2VA Nasal Mask | Total
Number analyzed (Participants) | 73 | 63 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 50 | 111
  >=65 years | 12 | 13 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 33 | 80
  Male | 26 | 30 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 73 | 63 | 136

OUTCOME MEASURES:

1. Primary Outcome: Time to First Intervention
Description: The time period between the beginning of standard of care propofol bolus and/or start of propofol infusion to time of initiation of the first intervention for airway management.
Time Frame: Usually 5 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Oxygen Via Nasal Cannula (Standard of Care) | Oxygen Via SuperNO2VA Nasal Mask
Number analyzed (Participants) | 73 | 63
minutes | 10 (12) | 19 (10)

2. Secondary Outcome: Number of Subjects Receiving Interventions for Airway Management
Description: Number of subjects receiving interventions for airway management including chin up and/or jaw thrust, oral and/or nasal airway insertion, mask ventilation, intubation with endotracheal tube (ETT) or laryngeal mask airway (LMA) insertion
Time Frame: Duration of colonoscopy procedure (usually 30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxygen Via Nasal Cannula (Standard of Care) | Oxygen Via SuperNO2VA Nasal Mask
Number analyzed (Participants) | 73 | 63
Participants | 46 | 14

3. Secondary Outcome: Duration of Intervention
Description: Duration of intervention
Time Frame: Duration of colonoscopy procedure (usually 30 minutes)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Oxygen Via Nasal Cannula (Standard of Care) | Oxygen Via SuperNO2VA Nasal Mask
Number analyzed (Participants) | 73 | 63
minutes | 19 (28) | 12 (31)

4. Secondary Outcome: Oxygen Saturation Reading- Median
Description: Oxygen saturation reading- Median
Time Frame: Duration of colonoscopy procedure (usually 30 minutes)
Measure: Median (Inter-Quartile Range); unit: percentage of oxygen saturation
Arm/Group | Oxygen Via Nasal Cannula (Standard of Care) | Oxygen Via SuperNO2VA Nasal Mask
Number analyzed (Participants) | 73 | 63
percentage of oxygen saturation
  Baseline | 100.0 [99 to 100] | 100 [99 to 100]
  2 minutes after induction | 98 [94 to 100] | 100 [99 to 100]
  4 minutes after induction | 99 [97 to 100] | 100 [99 to 100]
  6 minutes after induction | 99 [97 to 100] | 100 [99 to 100]
  5 minutes before end of procedure | 99 [97 to 100] | 100 [99 to 100]
  end of procedure | 98 [97 to 100] | 100 [99 to 100]

5. Secondary Outcome: Oxygen Saturation- Lowest Reading
Description: Oxygen saturation- Lowest reading
Time Frame: Duration of colonoscopy procedure (usually 30 minutes)
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Oxygen Via Nasal Cannula (Standard of Care) | Oxygen Via SuperNO2VA Nasal Mask
Number analyzed (Participants) | 73 | 63
percentage of oxygen saturation
  Baseline | 99.11 (1.76) | 99.23 (1.53)
  2 minutes after induction | 96.22 (6.12) | 99.31 (1.47)
  4 minutes after induction | 97.57 (4.79) | 99.39 (1.21)
  6 minutes after induction | 98.17 (3.32) | 99.52 (0.82)
  5 minutes before end of procedure | 97.76 (2.66) | 99.33 (1.03)
  end of procedure | 97.94 (2.11) | 99.19 (1.11)

6. Secondary Outcome: Number of Participants With Oxygen Saturation- Reading Below 90%
Description: Number of participants with oxygen saturation- reading below 90%
Time Frame: Duration of colonoscopy procedure (usually 30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxygen Via Nasal Cannula (Standard of Care) | Oxygen Via SuperNO2VA Nasal Mask
Number analyzed (Participants) | 73 | 63
Participants | 16 | 3

7. Secondary Outcome: Tidal Volume (VT)
Description: Tidal volume (VT) defined as the volume of air displaced between inhalation and exhalation.
Time Frame: Duration of colonoscopy procedure (usually 30 minutes)
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Oxygen Via Nasal Cannula (Standard of Care) | Oxygen Via SuperNO2VA Nasal Mask
Number analyzed (Participants) | 73 | 63
milliliters
  Baseline | 1032.80 (583.74) | 1011.39 (462.30)
  2 minutes after induction | 527.01 (367.54) | 625.31 (380.17)
  4 minutes after induction | 533.26 (467.47) | 589.22 (380.58)
  6 minutes after induction | 540.16 (417.28) | 613.15 (510.71)
  5 minutes before end of procedure | 610.38 (584.06) | 735.76 (614.42)
  end of procedure | 724.72 (538.90) | 879.52 (650.92)

8. Secondary Outcome: Respiratory Rate (RR)
Description: Respiratory Rate (RR)
Time Frame: Duration of colonoscopy procedure (usually 30 minutes)
Measure: Mean (Standard Deviation); unit: respiration per minute
Arm/Group | Oxygen Via Nasal Cannula (Standard of Care) | Oxygen Via SuperNO2VA Nasal Mask
Number analyzed (Participants) | 73 | 63
respiration per minute
  Baseline | 15.07 (4.57) | 15.36 (4.15)
  2 minutes after induction | 15.15 (5.32) | 15.21 (4.39)
  4 minutes after induction | 17.77 (5.36) | 16.95 (4.57)
  6 minutes after induction | 18.70 (4.87) | 17.48 (4.77)
  5 minutes before end of procedure | 18.39 (5.17) | 17.02 (4.40)
  end of procedure | 17.69 (4.5) | 17.50 (5.63)

9. Secondary Outcome: Minute Ventilation (MV)
Description: Minute ventilation (MV)
Time Frame: Duration of colonoscopy procedure (usually 30 minutes)
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | Oxygen Via Nasal Cannula (Standard of Care) | Oxygen Via SuperNO2VA Nasal Mask
Number analyzed (Participants) | 73 | 63
Liters per minute
  Baseline | 14.29 (8.01) | 14.52 (6.31)
  2 minutes after induction | 8.41 (6.44) | 9.16 (5.96)
  4 minutes after induction | 8.82 (6.86) | 9.62 (6.76)
  6 minutes after induction | 9.36 (5.99) | 9.94 (8.06)
  5 minutes before end of procedure | 10.29 (8.27) | 12.18 (10.82)
  end of procedure | 12.21 (9.19) | 13.48 (9.01)

ADVERSE EVENTS:
Time Frame: From the beginning of the study until discharge from the Post Anesthesia Recovery Room (Usually 2 hours)
Arm/Group | Oxygen Via Nasal Cannula (Standard of Care) | Oxygen Via SuperNO2VA Nasal Mask
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/70
Other Adverse Events (participants affected / at risk) | 0/79 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT03139448/Prot_SAP_000.pdf